CLINICAL TRIAL: NCT01602770
Title: Prospective, Non-interventional, 2-year Post-authorization Safety Study for QLAIRA®
Brief Title: Qlaira Post-authorization Safety Study Related to Most Common Adverse Events in Mexican Women Who Wish to Avoid Pregnancy
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16233; QL1210MX (Other: company internal)
Record Dates: First submitted 2012-05-18; First posted 2012-05-21 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Contraception
Keywords: Oral contraceptives; Adverse events; Safety profile; Contraceptive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Qlaira is taken daily continously with no pause between cycles in a four-phasic dose regimen, making up a treatment of up to 28 days. The first two tablets contain 3 mg Estradiol Valerate (E2V). The next five tablets include 2 mg E2V and 2 mg Dienogest (DNG) followed by 17 tablets with 2 mg E2V and 3 mg DNG. Finally, there are two tablets with 1 mg E2V and two placebo tablets.
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027) — Qlaira is taken daily continously with no pause between cycles in a four-phasic dose regimen, making up a treatment of up to 28 days. The first two tablets contain 3 mg Estradiol Valerate (E2V). The next five tablets include 2 mg E2V and 2 mg Dienogest (DNG) followed by 17 tablets with 2 mg E2V and 3 mg DNG. Finally, there are two tablets with 1 mg E2V and two placebo tablets.

SUMMARY:
Qlaira is a combined oral contraceptive (COC) containing dienogest/estradiol valerate being the first oral contraceptive delivering estradiol. It has been recently approved in Mexico. To evaluate the clinical profile of this drug combination under routine medical condition, a post-authorization safety study required by Mexican Health Authorities will be conducted in Mexican women.

The study will be performed as a descriptive study, no hypothesis will be tested. The cohort consists of 300 new users (first-ever users or switchers) of Qlaira under routine medical conditions. Subjects should provide all necessary information on health-related events or changes in health status during Qlaira use.

Primary variable will be the incidence of Adverse Events (AE) at any time point, whether or not related to Qlaira during at least 2 years of observation.

In order to comply with the criteria of a non-interventional study, women only will be informed about the study, asked to participate and included in the study after Qlaira has been prescribed.

Study patients follow-up will be done in accordance with common clinical practice as described at Mexican Official Guidelines for prescription of Family Planning Methods (NOM 005-SSA2-1993).

ELIGIBILITY:
Inclusion Criteria:

Healthy women of reproductive age who are:

* Seeking fertility control with oral contraception at least for one year
* Able to go back to medical office on regular basis

Exclusion Criteria:

Women with risk parameters of arterial or venous thrombotic diseases such as:

* Smoke, if over age 35
* Deep vein thrombosis or pulmonary embolism, now or in the past
* Cerebrovascular disease
* Coronary artery disease
* Thrombogenic valvular or thrombogenic rhythm diseases of the heart
* Inherited or acquired hypercoagulopathies
* Uncontrolled hypertension
* Diabetes with vascular disease
* Headaches with focal neurological symptoms or have migraine headaches with or without aura if over age 35
* Undiagnosed abnormal genital bleeding
* Breast cancer or other estrogen- or progestin-sensitive cancer, now or in the past
* Liver tumors, benign or malignant, or liver disease
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cohort of healthy women of reproductive age currently Qlaira users from selected obstetrics and gynecology (Ob/Gyn) primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events collection | After 24 months
Continuation rate, as proportion of patients still using Qlaira | After 24 months

SECONDARY OUTCOMES:
Reasons for discontinuation related or unrelated to adverse events | After 24 months
Patient satisfaction with Qlaira | After 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Mexico